CLINICAL TRIAL: NCT06126159
Title: MRI Functional Imaging Characteristics and Fat Quantification of CT-fat-free Renal Neoplasms: Relationships With Histological Classifications and Molecular Markers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li-Jen Wang, Medical Imaging Department Director, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201802271A3
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Kidney Neoplasms
Keywords: kidney; angiomyolipoma; renal cell carcinoma; imaging characteristics; magnetic resonance imaging; immunohistochemistry stain
MeSH Terms: conditions — Kidney Neoplasms; Angiomyolipoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multiparametric and fat-detection magnetic resonance imaging (MRI) (Experimental): detecting the small amount of fat with the use of fat-detecting pulse sequences on MRI
  Interventions: Diagnostic Test: multiparametric and fat-detection magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: multiparametric and fat-detection magnetic resonance imaging (MRI) — Differentiating of renal AMLs with minimal fat and RCCs

SUMMARY:
The knowledge of the histological diagnosis and its subtype of a renal parenchymal tumor is important for determine whether the choice of a specific regimen of chemotherapy, target therapy and immunotherapy could be suitable and effective for treating this tumor. Computed tomography (CT) has been considered as an excellent imaging modality for detecting intra-tumoral fat, and most of renal angiomyolipomas (AML) could be thus confidently diagnosed on computed tomography by showing intra-tumoral fat. However, if a renal parenchymal tumor has no detectable fat in the tumor on computed tomography, there is a long list of its diagnosis including benign neoplasms as angiomyolipoma with minimal fat, oncocytoma, metanephric adenoma, etc., epitheloid angiomyolipoma (eAML) malignant potential, malignant neoplasms as renal cell carcinoma (RCC), sarcoma, malignant eAML, etc. Furthermore, there are three kinds of anticancer drug (antiangiogenetic drug, mammalian target of rapamycin inhibitors, immune modulators, and whether the anticancer drug is effective mainly depending on subtypes of RCCs. Nonetheless, computed tomography could not reliably differentiate histological types of renal parenchymal masses except renal AMLs with abundant fat. Therefore, for patients without established diagnoses by imaging examinations, further biopsy of the renal tumor is usually mandatory to validate the histological diagnosis and subtype. Thus, this study plans to enroll 60 patients with renal parenchymal masses which show no intra-tumoral fat on computed tomography. All enrolled patients will undergo multiparametric and fat-detection magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Multiparametric MRI includes not only conventional T1-weighted and T2-weighted images but also diffusion weighted images and dynamic contrast enhanced images. Fat-detection MRI include fat-suppressed images by frequency selection, out-of-phase images (compared with in-phase image) and fat quantification pulse sequence for determining the presence or absence of intra-tumoral fat as well as measuring fat amount. We will record MRI characteristics of the renal parenchymal tumors of the patients. If the patients undergo further biopsy for establishing histological diagnoses and subtypes after MRI examination, the specimens of the renal tumor obtained from biopsy will be further analyzed by immunohistochemistry stain (IHC), quantitative real-time polymerase chain reaction (qPCR) and western blot after obtainment of the patient's informed consent. The MRI characteristics of the renal parenchymal tumors of the patients will be then correlated with histological examination, IHC, qPCR and western blot examinations of the tumors. We will then use univariate and multivariate analyses to determine whether MRI characteristics are useful as imaging surrogates for predicting biomarkers as histological diagnosis, subtypes, IHC, qPCR and western blot results.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years old
2. Have renal parenchymal masses with no detectable intra-tumoral fat on computed tomography (CT)
3. Normal renal function (i.e.: estimated glomerular filtration rate ≧ 60 mL/min/1.73 m2)
4. No allergy history of iodinated contrast medium

Exclusion Criteria:

1. Pregnant or lactating woman
2. Withdrawal of informed consent
3. Those who have not completed MRI
4. Those who did not receive renal tumor biopsy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MR characteristics assessment- T2WI | 3 years
  T2-weighted images (T2WI)
MR characteristics assessment- ADC | 3 years
  Apparent diffusion coefficient (ADC)
MR characteristics assessment- IVIM | 3 years
  Intravoxel incoherent motion (IVIM)

SECONDARY OUTCOMES:
Immunohistochemistry (IHC) statin- mTOR | 3 years
  The IHC stains for protein reactions of total mTOR are analyzed using electronic files obtained from Aperio Digital pathology slide Scanner.
Immunohistochemistry (IHC) statin- Phospho-mTOR | 3 years
  The IHC stains for protein reactions of Phospho-mTOR (pmTOR) are analyzed using electronic files obtained from Aperio Digital pathology slide Scanner.
Immunohistochemistry (IHC) statin- Rheb | 3 years
  The IHC stains for protein reactions of Rheb are analyzed using electronic files obtained from Aperio Digital pathology slide Scanner.
Immunohistochemistry (IHC) statin- S6K | 3 years
  The IHC stains for protein reactions of S6K are analyzed using electronic files obtained from Aperio Digital pathology slide Scanner.
Immunohistochemistry (IHC) statin- pS6K | 3 years
  The IHC stains for protein reactions of pS6K are analyzed using electronic files obtained from Aperio Digital pathology slide Scanner.
Quantitative Real-Time polymerase chain reaction (qPCR) | 3 years
  We extract RNA from tumor cells using RNeasy Mini Kit (Qiagen), according to the manufacturer's protocol and reverse transcription of RNA into cDNA is done using with PrimeScript TM RT reagent kit (Takara Bio Inc.), followed by amplified by polymerase chain reaction (PCR) using the SYBR Green SuperMix (BioRad, Hercules, CA).
  The quantitative real-time PCR (qPCR) test including primer sequences of the PI3K/AKT/mTOR pathway genes including Phosphatase and tensin homolog (PTEN), mTOR, ribosomal protein S6 kinase B1 (S6K1), Ras Homolog, MTORC1 Binding (RHEB) and Eukaryotic translation initiation factor 4E-binding protein 1 (4EBP1) genes are analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jen Wang, M.D., M.P.H., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Li-Jen Wang, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Plan to make individual participant data